CLINICAL TRIAL: NCT03480022
Title: A Randomized Placebo-controlled Double Blind Trial of Liraglutide 3 mg [Saxenda] on Weight, Body Composition, Hormonal and Metabolic Parameters in Obese Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Liraglutide 3mg (Saxenda) on Weight, Body Composition, Hormonal and Metabolic Parameters in Obese Women With PCOS
Acronym: SAXAPCOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Scientific Director of Research, Woman's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1198-4126
Record Dates: First submitted 2018-03-13; First posted 2018-03-27 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Pre Diabetes; Polycystic Ovary Syndrome; Obesity Android
Keywords: prediabetes; PCOS; GLP-1 agonist; weight loss
MeSH Terms: conditions — Glucose Intolerance; Polycystic Ovary Syndrome; Obesity, Abdominal; Prediabetic State; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double- Blind 2:1 Drug: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide Pen Injector (Saxenda) (Experimental): Start injection liraglutide 0.6 mg subcutaneously (SC) 1week daily (QD), step up to 1.2 mg SC QD for 1week, to 1.8 mg SC QD for 1 week, 2.4 mg SC QD for 1week, to a final dose of 3.0 mg liraglutide SQ daily
  Interventions: Drug: Liraglutide Pen Injector [Saxenda]
- Placebo liraglutide pen injector (Placebo Comparator): Start injection of placebo liraglutide 0.6 mg subcutaneously (SC) 1week daily (QD), step up to 1.2 mg SC QD for 1week, to 1.8 mg SC QD for 1 week, 2.4 mg SC QD for 1week, to a final dose of 3.0 mg placebo liraglutide SQ daily
  Interventions: Drug: Placebo Liraglutide Pen Injector

INTERVENTIONS:
Drug: Liraglutide Pen Injector [Saxenda] — daily sc injection of liraglutide with final dose of 3mg daily
  Other Names: Liraglutide 3mg; Saxenda
  Arms: Liraglutide Pen Injector (Saxenda)
Drug: Placebo Liraglutide Pen Injector — daily sc injection of placebo liraglutide with final dose of 3mg daily of placebo
  Other Names: Placebo Saxenda; Placebo liraglutide 3 mg
  Arms: Placebo liraglutide pen injector

SUMMARY:
There is a growing need to develop pharmacologic interventions to improve metabolic function in women with polycystic ovary syndrome (PCOS). Given that PCOS is a frequent condition and weight loss is essential but difficult to achieve, it is important to study if the effect on body weight reported in other studies can be confirmed in a selected population of hyperandrogenic patients, especially with medications currently approved for weight reduction. High dose liraglutide alone results in significant weight reduction in obese women without PCOS. There is limited data on weight loss with high dose liraglutide in non-diabetic females with PCOS treated with this agent . Studies on the effect of anti-obesity medication combined with lifestyle changes on body weight and composition and androgen excess in obese women diagnosed with PCOS are lacking. The investigators aim to elucidate the most efficacious weight reduction regime in obese PCOS women. The investigators further hope to determine which treatment(s) addressing the multifaceted disturbances of this disorder in patients with PCOS and obesity emerges as the preferable therapy.

DETAILED DESCRIPTION:
The drug, liraglutide 3.0 mg was approved for chronic weight management in management in obese adults with an initial BMI of 30 kg/m2 or greater or in overweight adults BMI of 27 kg/m2 or greater with at least one weight-related co-morbid condition as an adjunct to a reduced-calorie diet and increased physical activity. Liraglutide is an acylated human glucagon-like peptide -1 (GLP-1) analog that binds to and activates the GLP-1 receptor. It lowers body weight through decreased caloric intake while stimulating insulin secretion and reducing glucagon via a glucose-dependent mechanism. For obesity management, patients may lose weight with GLP-1 receptor agonists due to other unique actions. Glucagon-like peptide-1 receptor agonists (GLP-1RAs) can slow gastric emptying and increase satiety. While predictors of weight loss success for the general population are available (protein intake, weight loss medications), predictors of weight loss success may differ between normal and hyperandrogenic women. Glucagon-like peptide 1 agonists are linked with dose dependent weight lowering potential in different obesity related populations. The weight loss effects of GLP-1RAs previously demonstrated in diabetic and obese non-diabetic patients, offer a unique opportunity to expand the medical options available to patients with PCOS.

Given this lack of information, the aim of the present study was to investigate the effects of liraglutide 3mg vs. placebo on body composition as well as hormonal and metabolic features in non-diabetic obese women with PCOS.The non-diabetic obese female with PCOS offers a unique model to study the relationship between insulin resistance and adiposity. The investigators propose a double-blind, placebo-controlled 30-week trial designed to directly examine the therapeutic effects of liraglutide 3 mg (LIRA 3 mg) compared to placebo on body weight, hormonal and cardiometabolic parameters in obese non-diabetic women with PCOS. All patients will receive diet and lifestyle counseling, including advice on exercise commencing during the lead-in period and continuing throughout the study. In this study, the investigators will examine the efficacy of LIRA 3mg on body weight and body composition, reproductive function metabolic parameters and cardiovascular risk factors in a well-defined group of pre-menopausal obese non-diabetic women with hyperandrogenism, focusing on the relationship to obesity and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* 18-45 years of age
* BMI ≥30 kg/m2 or BMI ≥27 kg/m2 with one or more obesity-associated co-morbid conditions (e.g. hypertension, and dyslipidemia)
* PCOS- NIH criteria hyperandrogenism and irregular menstrual cyclicity
* Non-diabetic as determined by a 75 gram oral glucose tolerance test (OGTT) and hemoglobin A1C. Non-diabetic is inclusive of women with impaired fasting glucose (IFG), impaired glucose tolerance (IGT), or both (IFG/IGT). Participants with diabetes will be excluded
* Willing to use effective contraception consistently during therapy which is defined as:

  * an intrauterine device, tubal sterilization, or male partner vasectomy, or
  * combination of two barrier methods with one being male condom.
* Written consent for participation in the study

Exclusion Criteria:

* Presence of significant systemic disease, cerebrovascular disease, clinically significant cardiac abnormalities or heart problems including congestive heart failure, unstable angina or acute myocardial infarction, current infectious liver disease, acute stroke or transient ischemic attacks, history of pancreatitis, or diabetes mellitus (Type 1 or 2)
* Any hepatic diseases in the past (infectious liver disease, viral hepatitis, toxic hepatic damage, jaundice of unknown etiology) or severe hepatic insufficiency and/or significant abnormal liver function tests defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
* Renal impairment (e.g., serum creatinine levels ≥1.4 mg/dL for women, or eGFR <60 mL/min/1.73 m2) or history of unstable or rapidly progressing renal disease or end stage renal disease.
* Uncontrolled thyroid disease (documented normal TSH), Cushing's syndrome, congenital adrenal hyperplasia or clinically significant elevations in prolactin levels. The clinical significance of prolactin levels will be determined by the treating physician
* Significantly elevated triglyceride levels (fasting triglyceride > 400 mg %)
* Untreated or poorly controlled hypertension (sitting blood pressure > 160/95 mm Hg)
* Use of hormonal medications, the use of medications that cause clinically significant weight gain or loss (prescription or OTC) and medications known to exacerbate glucose tolerance (such as isotretinoin, hormonal contraceptives, GnRH analogues, glucocorticoids, anabolic steroids, C-19 progestins) including herbal medicines for at least 8 weeks. Use of anti-androgens that act peripherally to reduce hirsutism such as 5-alpha reductase inhibitors (finasteride, spironolactone, flutamide) for at least 4 weeks
* Prior history of a malignant disease requiring chemotherapy
* Family or personal history of familial medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Known hypersensitivity or contraindications to use GLP1 receptor agonists
* Use of metformin, thiazolidinediones, GLP-1 receptor agonists, dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium/glucose co-transporter 2 (SGLT2) inhibitors or weight loss medications (prescription or OTC) stopped for at least 4 weeks
* Prior use of medication to treat diabetes except gestational diabetes
* Eating disorders (anorexia, bulimia) or gastrointestinal disorders
* Suspected pregnancy (documented negative serum pregnancy test), desiring pregnancy in next 15 months, breastfeeding, or known pregnancy in last three months
* Active or prior history of substance abuse (smoke or tobacco use within past 6 months) or significant intake of alcohol
* Previous bariatric surgery or device intervention for obesity
* Patient not willing to use barrier contraception during study period (unless sterilized or have an IUD)
* History of major depressive or other severe psychiatric disorders
* Inability or refusal to comply with protocol
* Currently participating or having participated in an experimental drug study in previous three months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients must be female to have the disorder being studied since it involved the female reproductive system
Enrollment: 88 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Dean, PharmD, Study Chair — Woman's Hospital Foundation IRB
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elkind-Hirsch KE, Chappell N, Shaler D, Storment J, Bellanger D. Liraglutide 3 mg on weight, body composition, and hormonal and metabolic parameters in women with obesity and polycystic ovary syndrome: a randomized placebo-controlled-phase 3 study. Fertil Steril. 2022 Aug;118(2):371-381. doi: 10.1016/j.fertnstert.2022.04.027. Epub 2022 Jun 13. PMID 35710599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 88 recruited, 82 met criteria and randomized Six excluded after consenting
Period: Overall Study
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Started | 55 | 27
Completed | 44 | 23
Not Completed | 11 | 4
Not completed — Pregnancy | 2 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Medication concerns | 1 | 0
Not completed — Family member COVID exposure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector | Total
Number analyzed (Participants) | 55 | 27 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (6) | 31.8 (5.6) | 31.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 27 | 82
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 9 | 22
  White | 42 | 18 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 27 | 82
Body mass Index [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated as kg/meters squared
  kg/m^2 | 42 (6.7) | 43.9 (7.5) | 42.4 (7)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Body Weight (BW)
Description: Treatment impact on change in body weight after 32 weeks of treatment.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: kilogram
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
kilogram | 104.7 (2.9) | 117.9 (5)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; Repeated measures general linear model (SS/drug treatments by visits) where arm of drug therapy as between subjects effect and visit (baseline and 32 weeks of treatment) as within subject effect; Test type: Superiority; p < 0.002, ANOVA; Nested repeated measures design

2. Primary Outcome: Free Androgen Index (FAI)
Description: Drug treatment effect on free androgen levels as calculated as FAI= total testosterone (T) concentrations divided by sex hormone binding globulin (SHBG) levels. A higher score indicates a worse outcome (more androgenic).
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
index score | 5.98 (0.6) | 6.4 (.75)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.006, ANOVA; Nested repeated measures design

3. Secondary Outcome: Body Mass Index (BMI)
Description: Treatment effect in reducing body mass
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: kilogram/meter squared
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
kilogram/meter squared | 39.1 (1.1) | 43.4 (1.8)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANOVA; Repeated measures nested design

4. Secondary Outcome: Change in Percent Body Weight
Description: Treatment effect on reducing body weight expressed as percent body weight loss from baseline
Time Frame: Change from baseline (time 0) to study end (32 weeks)
Measure: Mean (Standard Error); unit: percentage loss in body weight
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
percentage loss in body weight | 5.7 (0.75) | 1.4 (1.09)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; Test type: Superiority; p < 0.002, ANOVA; one-way ANOVA

5. Secondary Outcome: 5% Weight Loss From Baseline
Description: Frequency of patients achieving 5% weight loss from baseline with treatment
Time Frame: 32 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
Participants | 25 | 5
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; Test type: Superiority; p < 0.007, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: 10% Body Weight Loss From Baseline
Description: Frequency of patients with at least 10% reduction in body weight from baseline
Time Frame: 32 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
Participants | 13 | 2
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; Test type: Superiority; p < 0.049, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Abdominal Adiposity (Waist Circumference [WC]
Description: Treatment effect on loss of WC (abdominal adiposity) with drug treatment
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
centimeters | 100.9 (2.0) | 109.9 (3.3)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.011, ANOVA; Nested repeated measures design

8. Secondary Outcome: Waist-to-Hip Ratio
Description: Change in central adiposity with treatment as measured by WHR. A reduction in ratio indicates a decrease in truncal fat.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
ratio | 0.81 (0.009) | 0.85 (0.015)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.038, ANOVA; Nested repeated measures design

9. Secondary Outcome: Waist-to Height Ratio [WHtR])
Description: Treatment effect on loss of central adiposity as determined by WHt ratio. The lower the ratio indicates less abdominal adiposity.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
ratio | 0.62 (0.014) | 0.67 (0.02)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.048, ANOVA; Nested repeated measures design

10. Secondary Outcome: Total Fat Mass Evaluated by DEXA
Description: Treatment effect on reduction of fat mass (kg)
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: kilogram
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
kilogram | 49.3 (2.1) | 56.8 (3.3)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.018, ANOVA; Nested repeated measures design

11. Secondary Outcome: Total Body Fat (%) by DXA
Description: Treatment effect on reduction of percent body fat by DXA
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: percent fat mass
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
percent fat mass | 46.0 (0.9) | 47.9 (0.96)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.028, ANOVA; Nested repeated measures design

12. Secondary Outcome: Android-Gynoid Ratio (AGR) by DXA
Description: Treatment impact on AGR, measure of central adiposity, as determined by DXA. A lower AGR indicates a reduction in central adiposity.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
ratio | 1.05 (0.01) | 1.08 (0.03)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.034, ANOVA; Nested repeated measures design

13. Secondary Outcome: Trunk/Leg Fat Ratio (TLR) by DXA
Description: Treatment impact on TLR after 32 weeks. A reduction in TLR indicates a loss of central fat.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
ratio | 1.02 (0.03) | 1.07 (0.04)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.035, ANOVA; Nested repeated measures design

14. Secondary Outcome: Menstrual Cycle Frequency
Description: Drug treatment impact on normalization of cycle frequency (cycle every 28-30 days). All cycle data is expressed as number of menses annualized to one year.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: menses per year
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
menses per year | 8.65 (0.4) | 4.8 (0.65)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Nested repeated measures design

15. Secondary Outcome: Total Testosterone Concentrations (T)
Description: Drug treatment effect on total testosterone concentrations
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
ng/dL | 45.4 (3.0) | 46.8 (4.1)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, ANOVA; Nested repeated measures design

16. Secondary Outcome: Adrenal Dehydroepiandrosterone Sulfate (DHEAS)
Description: Treatment efficacy in reducing adrenal hyperandrogenism
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mcg/dL
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mcg/dL | 177.1 (14.2) | 171.3 (16.8)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, ANOVA; Nested repeated measures design

17. Secondary Outcome: Fasting Blood Glucose (FG)
Description: Treatment effect on fasting glucose prior to an oral glucose tolerance test (OGTT)
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mg/dL | 90.2 (1.3) | 94.3 (2.2)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.021, ANOVA; Nested repeated measures design

18. Secondary Outcome: OGTT Mean Blood Glucose (MBG)
Description: Treatment effect on MBG measured during the oral glucose tolerance test. A decrease in MBG shows improvement in glycemia.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mg/dL | 109.4 (2.9) | 125.5 (4.8)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.009, ANOVA; Nested repeated measures design

19. Secondary Outcome: Fasting Insulin Sensitivity (HOMA-IR)
Description: Treatment effect on the HOMA-IR which is an insulin resistance measured derived from fasting blood glucose and insulin . The higher the number the more insulin resistant.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
index score | 4.1 (0.6) | 5.2 (1.1)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.035, ANOVA; Nested repeated measures design

20. Secondary Outcome: Matsuda Insulin Sensitivity Index Derived From the OGTT (SI OGTT)
Description: The SI OGTT is a measure of peripheral insulin sensitivity derived from the insulin and glucoses measured during an OGTT. A increase in SI OGTTindicates greater insulin sensitivity
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
index score | 3.7 (0.43) | 3.0 (0.48)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.028, ANOVA; Nested repeated measures design

21. Secondary Outcome: Corrected First Phase Insulin Secretion (IGI/HOMA-IR)
Description: Treatment effect on insulin secretion from 0 to 30 minutes after glucose load corrected for by fasting insulin sensitivity. A higher score shows improved first phase insulin secretion in response to glucose.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
index score | 1.01 (0.18) | 0.8 (0.16)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.042, ANOVA; Nested repeated measures design

22. Secondary Outcome: Insulin Secretion- Insulin Sensitivity Index (Oral Disposition Index-IS-SI)
Description: Treatment effect on an estimation of Beta cell compensatory function, the IS-SI is derived by applying the concept of the disposition index to measurements obtained during the 2 hour OGTT and calculated as the index of insulin secretion factored by insulin sensitivity. A higher score shows improved pancreatic beta cell function relative to insulin sensitivity.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
index score | 532 (91) | 416 (69.7)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.033, ANOVA; Nested repeated measures design

23. Secondary Outcome: Total Cholesterol Levels
Description: Treatment impact on improving total cholesterol levels
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mg/dL | 176 (5.3) | 178 (8.8)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, ANOVA; Nested repeated measures design

24. Secondary Outcome: High Density Lipoprotein Cholesterol (HDL-C)
Description: Impact of treatment on HDL levels after 32 weeks of treatment
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mg/dL | 41 (1.8) | 42 (2.3)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, ANOVA; Nested repeated measures design

25. Secondary Outcome: Triglyceride Levels (TRG)
Description: Drug effect of TRG levels after treatment
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mg/dL | 109 (7.7) | 114 (11)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.016, ANOVA; Nested repeated measures design

26. Secondary Outcome: Triglyceride to HDL-Cholesterol Ratio (TRG/HDL-C)
Description: Treatment impact on TRG/HDL-C ratio which is a simple measure to estimate insulin action. A decrease in ratio indicates improvement in insulin sensitivity.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
ratio | 2.9 (0.26) | 3.0 (0.45)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.028, ANOVA; Nested repeated measures design

27. Secondary Outcome: Triglyceride and Glucose Index (TyG)
Description: Treatment impact on the TyG index which estimates insulin resistance. A reduction in TyG indicates an improvement in insulin action.
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: index score
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
index score | 8.39 (0.07) | 8.5 (0.09)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, ANOVA; Nested repeated measures design

28. Secondary Outcome: Systolic Blood Pressure
Description: Treatment impact on systolic blood pressure
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mmHg | 116.8 (2.7) | 123.3 (2.4)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, ANOVA; Nested repeated measures design

29. Secondary Outcome: Diastolic Blood Pressure (BP)
Description: Treatment impact on reducing diastolic blood pressure
Time Frame: 32 weeks of treatment
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
Number analyzed (Participants) | 44 | 23
mmHg | 77.6 (1.6) | 78.1 (1.3)
Statistical Analysis 1: Comparison: Liraglutide Pen Injector (Saxenda) vs Placebo Liraglutide Pen Injector; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, ANOVA; Nested repeated measures design

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Liraglutide Pen Injector (Saxenda) | Placebo Liraglutide Pen Injector
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/27
Other Adverse Events (participants affected / at risk) | 40/55 | 8/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liraglutide Pen Injector (Saxenda) (N=55) | Placebo Liraglutide Pen Injector (N=27)
Nausea (Gastrointestinal disorders) | 14 | 3
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Heartburn (Gastrointestinal disorders) | 2 | 1
Reflux (Gastrointestinal disorders) | 2 | 0
Indigestion (Gastrointestinal disorders) | 2 | 0
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 | 0
prolonged menstrual bleeding (Reproductive system and breast disorders) | 3 | 1
no menses (Reproductive system and breast disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03480022/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03480022/ICF_000.pdf